CLINICAL TRIAL: NCT06141343
Title: Project V - A Randomized Controlled Prospective Study of the Next-generation Probiotic, Veillonella Atypica FB0054, vs Placebo in Healthy Adults
Brief Title: A Study of the Next-generation Probiotic, Veillonella Atypica FB0054 vs Placebo
Acronym: ProjectV
Status: Completed | Type: Observational
Sponsor: FitBiomics, Inc. (Industry)
Collaborators: People Science, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FB004
Record Dates: First submitted 2023-08-03; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Veillonella atypica FB0054: Active ingredient dietary supplement group
  Interventions: Dietary Supplement: Veillonella atypica FB0054
- Placebo: No active ingredient
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Veillonella atypica FB0054 — Veillonella contains Veillonella atypica FB0054 as the active ingredient with microcrystalline cellulose and hypromellose as excipients. The two doses are 15 billion cfu (high dose) and 7.5 billion cfu (low dose). Placebo capsules contain microcrystalline cellulose and hypromellose. Both Veillonella and placebo are encapsulated in acid-resistant capsules to improve delivery to the large intestine, which participants will take orally at home on a daily basis for four weeks.
  Groups: Veillonella atypica FB0054
Other: Placebo — Placebo will be given as the non-active study control
  Groups: Placebo

SUMMARY:
In this study, the investigators are assessing the ability of Veillonella (Veillonella atypica FB0054) to decrease fatigue and increase energy in a heterogeneous cohort of healthy adults compared to placebo. Study subjects will fill out a baseline health and habit survey followed by daily and weekly surveys over a two week baseline period to understand their baseline habits, fatigue, and energy levels. After this, subjects will take one daily capsule orally of one of two doses of Veillonella or placebo for four weeks, while again filling out both daily and weekly surveys. Finally, there will be a two week washout period with no supplementation but only daily and weekly surveys. At the end of the study, there will be a final experience survey.

DETAILED DESCRIPTION:
Veillonella is a novel probiotic that can metabolize lactic acid into propionate, which is an energy source for the body. In previous research, the investigators have shown that Veillonella can improve endurance compared to placebo. In mouse studies, those mice who supplemented with V. atypica ran 13% longer in a run-to-exhaustion test than those mice who were given placebo. Furthermore, in a randomized controlled crossover pilot study, the investigators could show that Veillonella prevented 78.7% of the performance decline observed in the placebo group in a run-to-exhaustion model. The investigators have also conducted experiments that have resulted in this product being deemed Generally Regarded As Safe (GRAS).

Therefore, the investigators believe the Veillonella is safe and likely to provide significant benefits in terms of improved endurance, increased energy, and decreased fatigue. This research study is designed to test that hypothesis. FitBiomics is sponsoring this study to confirm these effects in a broader population. FitBiomics is the first company to develop this type of bacteria as a probiotic, and this will be the largest study testing the safety and efficacy of this probiotic.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged 18 - 65 years.
* Willing and able to provide written informed consent.
* Ability of the participant to comprehend the full nature and purpose of the study including possible risks and side effects.
* Agreement to comply with the protocol and study restrictions.
* Fluent in written and spoken English.
* In good general health as judged by the Investigator based on medical history.
* Willing to maintain daily exercise and diet habits throughout the 8 week study without making major lifestyle changes.
* Ability to use a personal smartphone device and download the Chloe app by People Science

Exclusion Criteria:

* Currently pregnant, planning to become pregnant, or lactating during the next 12 weeks
* Have a significant acute or chronic coexisting illness, disorder, or condition that contraindicates, in the Principal Investigator's judgment, entry to the study.
* Currently taking immunosuppressive medications.
* Is considered immunosuppressed for any reason.
* Currently taking medications that could impair the integrity of the gut epithelia
* Has symptoms or an illness, disorder, or cognition that impairs the integrity of the gut epithelia.
* Current antibiotic use or planned oral antibiotic use over the course of the study.
* Investigator believes that the participant may be uncooperative and/or noncompliant and should therefore not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in this study will be healthy adults interested in using Veillonella to reduce fatigue and increase energy. Subjects will be excluded from the study if they have conditions, diseases, or medications that could result in increased likelihood of AEs related to Veillonella use.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Changes in reported physical fatigue | 8 weeks
  The majority of primary endpoints for this study are questions on the survey which consist of rating scales (generally 1-5 or 1-9). Significant differences between groups for these endpoints will be assessed using an independent T test or Mann-Whitney U test depending on the observed distribution of the data. For significant changes over time within the same group, a dependent T test will be used.
Change in mental / emotional fatigue | 8 weeks
  The majority of primary endpoints for this study are questions on the survey which consist of rating scales (generally 1-5 or 1-9). Significant differences between groups for these endpoints will be assessed using an independent T test or Mann-Whitney U test depending on the observed distribution of the data. For significant changes over time within the same group, a dependent T test will be used.
Change in Multi-dimensional Fatigue Inventory Questionnaire | 8 weeks
  The majority of primary endpoints for this study are questions on the survey which consist of rating scales (generally 1-5 or 1-9). Significant differences between groups for these endpoints will be assessed using an independent T test or Mann-Whitney U test depending on the observed distribution of the data. For significant changes over time within the same group, a dependent T test will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Scheiman, PhD, Principal Investigator — FitBiomics, Inc.
Locations (1):
- FitBiomics, Inc., New York, New York, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT06141343/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT06141343/ICF_001.pdf